CLINICAL TRIAL: NCT04845854
Title: Prevalence of Oral Side Effects Associated With Chemo and Radiotherapy for Treating Head and Neck Cancer: a Cross-sectional Study
Brief Title: Prevalence of Oral Side Effects Associated With Chemo and Radiotherapy for Treating Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dalia Mohamed abo el -fadel, post graduation student, Cairo University
Other Study IDs: 4221
Record Dates: First submitted 2021-04-07; First posted 2021-04-15 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2021-04

CONDITIONS: Oral Complications of Chemotherapy and Head and Neck Radiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

SUMMARY:
A cross-sectional study will be conducted to report oral complications during chemo and radiotherapy treatment in case of patients diagnosed with head and neck cancer and the effect of theses oral side effects on patients' quality of life which will in turn allow the implication of preventive measures

DETAILED DESCRIPTION:
the primary out come of this study is to report oral side effects associated with chemo and radiotherapy used for treating head and neck cancer .patient will be enrolled and data will be collected from the national institute of cancer in Egypt. this will be done through filling the modified ( Edmonton Symptom Assessment System) ESAS questionnaire used to asses different oral side effects in cancer patients. history taking and Clinical examination will be done for each patient enrolled in the study after obtaining their consent form by the main investigator. each and every oral manifestations will be measured by a specific scale . the secondary outcome is identified as the assessment of the effect of oral complications on patients' quality of life which will be determined through completing UW-QOL(University of Washington-Quality Of Life) questionnaire version 4.during the study, patient , treatment and tumor variable will be considered and documented .Data collected form the patient and or from medical records will be saved and tabulated on computer for back up and finally statistically analyzed. A power analysis was designed to have adequate power to apply a statistical test of the research question regarding the degree to which oral adverse events can prevail among patients receiving chemotherapy or radiotherapy. According to the results of Minhas, Sadia, et al. -in which prevalence of oral adverse events was (92.6%)- and by adopting a confidence interval of (95%), a margin of error of (3%) with finite population correction; the predicted sample size (n) was a total of (292) cases. Sample size calculation was performed using Epi info for windows version 7.2

ELIGIBILITY:
Inclusion Criteria:

* Patients after the first week of their treatment till the end of their treatment protocol and at their follow-up visits
* patients who completed ESAS questioner
* Male and female patients from 20 -70 years old who are diagnosed with head and neck cancer.

Exclusion Criteria:

* Patients who didn't start their treatment before the examination
* Patients who refuse to participate in the study.
* Patients with leukemia or blood cell cancers, infants and children

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients who are diagnosed with head and neck cancer and started their chemo and radiotherapy treatment
Sampling Method: Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-09-03 (Actual)

PRIMARY OUTCOMES:
by ESAS questionnaire ,clinical examination of the patient | through study completion, an average of 1 year
  questionnaire is answered by the patient
oral mucositis assessed by WHO(world Health Organization) scale, clinical examination | through study completion, an average of 1 year
  grade(A)none , (I)mild ,(II)moderate (III)severe and( life threatening (B) 1 asymptomatic or mild pain,2moderate,3 severe,4 life threatening
xerostomia by CODs (Clinical oral dryness scale) | through study completion, an average of 1 year
  questionnaire completed with added clinical examination scored from 1-3indicate mild dryness then 4-6 moderate dryness and 8-10 severe dryness
dysphagia by VHNSS Version 2.0 (Vanderbilt Head and Neck Cancer Symptom Survey) | through study completion, an average of 1 year
  assess the severity of dysphagia by a questionnaire related to struggle during swallowing ,xerostomia, nutrition deficiency ,mucous secretion or taste changes ,mucositis and speech affection each scored from 0 (none) to 10 (severe).
pain assessed by numerical rating scale(NRS) | through study completion, an average of 1 year
  from 0 indicating no pain to 10 being worst pain

SECONDARY OUTCOMES:
quality of life assessment QOL-Version 4(Washington University Quality Of Life ) questionnaire | through study completion, an average of 1 year
  questionnaire consists of 12 single question domains, these having between 3 and 6 response options that are scaled evenly from 0 (worst) to 100 (best) according to the hierarchy of response.
  The domains are pain, appearance, activity, recreation, swallowing, chewing, speech, shoulder, taste, saliva, mood and anxiety

CONTACTS AND LOCATIONS:
Overall Officials: dalia m abo el fadel, master, Principal Investigator — dentist at hospital specialized centers
Locations (1):
- National Institute of Cancer in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No